CLINICAL TRIAL: NCT04654767
Title: Inflammatory Profiling in Chronic Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Lung Vascular Research (Other)
Collaborators: Medical University of Graz (Other); Medical University of Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: LBILVR-KLI 884-B
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Hypertension
Keywords: Vascular Diseases; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Hypertension, Pulmonary; Vascular Diseases; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, explant lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD-PH group: Patients with confirmed COPD and pulmonary hypertension
  Interventions: Other: Tissue sampling
- IPF-PH: Patients with confirmed pulmonary fibrosis and pulmonary hypertension
  Interventions: Other: Tissue sampling
- Control group: Control group without diagnosed COPD, IPF, or pulmonary hypertension
  Interventions: Other: Tissue sampling

INTERVENTIONS:
Other: Tissue sampling — Blood collection via venipuncture into citrate- or ethylenediaminetetraacetic (EDTA)-containing vacutainer tubes and into serum tubes. Explant lung tissue obtained from patients that underwent lung transplantation.
  Non-transplanted donor lungs that had been harvested for transplantation, but not implanted because of size-reduction serve as controls.

SUMMARY:
The aim of this study is to investigate the underlying inflammatory profile in patients with chronic lung disease and determine the association pulmonary hypertension.

DETAILED DESCRIPTION:
Chronic lung diseases (CLD), such as chronic obstructive pulmonary disease (COPD) and idiopathic pulmonary fibrosis (IPF) are often complicated by the presence of pulmonary hypertension (PH), where even a mild elevation of blood pressure in the pulmonary arteries is associated with an even poorer prognosis. In this study, we will investigate whether similarities exist in the inflammatory profile that could potentially underlie all forms of pulmonary hypertension. Inflammatory data will be generated using flow cytometry, expression profiling and histological analysis and compared to the associated clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung transplant with COPD or IPF, with associated PH
* Signed informed consent

Exclusion Criteria:

* patients without written informed consent
* Signs of any infection such as pneumonia, pulmonary tuberculosis or infections with pleural effusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing lung transplantation at the Medical University of Vienna
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of inflammatory cell profile | within 36 months
  The number of leukocytes (CD45+ cells) and derivatives (percentage lymphocytes, monocytes and neutrophils) will be measured by flow cytometry in explanted lung tissue and blood of patients with CLD-PH and controls.
  Values will be reported as %CD45+ and %total cells.

SECONDARY OUTCOMES:
Degree of pulmonary vascular disease | within 36 months
  Pulmonary vascular disease will be assessed by associated clinical data (mPAP (mmHg), PVR (WU))
  1. CLD without PH (mPAP <21 mmHg, or mPAP 21-24 mmHg with pulmonary vascular resistance (PVR) <3 Wood Units (WU)).
  2. CLD with PH (mPAP 21-24 mmHg with PVR ≥3 WU, or mPAP 25-34 mmHg) (CLD-PH).
  3. CLD with severe PH (mPAP ≥35 mmHg, or mPAP ≥25 mmHg with low cardiac index (<2.0 L·min-1·m-2)) (CLD-severe PH).

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Marsh, Principal Investigator — Ludwig Boltzmann Institute for Lung Vascular Research
Locations (1):
- Division of Thoracic Surgery, Department of Surgery, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided